CLINICAL TRIAL: NCT00781339
Title: A Phase IIa Open Label Study to Evaluate the Safety and Antimicrobial Effects of NVC-422 on Bacteriuria in Chronically Catheterized Subjects
Brief Title: Safety and Efficacy Study of NVC-422 on Bacteriuria in Catheterized Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NovaBay Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL0803; H-23765
Record Dates: First submitted 2008-10-28; First posted 2008-10-29 (Estimated); Last update posted 2011-09-12 (Estimated); Status verified 2011-09

CONDITIONS: Asymptomatic Bacteriuria
Keywords: Bacteriuria; Catheterized; Chronically Catheterized
MeSH Terms: conditions — Bacteriuria | interventions — NVC-422

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Active (Experimental)
  Interventions: Drug: sodium 2-(dichloroamino)-2-methylpropane-1-sulfonate monohydrate

INTERVENTIONS:
Drug: sodium 2-(dichloroamino)-2-methylpropane-1-sulfonate monohydrate — 0.1% NVC-422 in saline, up to 100 mL, Study Part 1 - once on Day 1 held in the bladder for 1 hour; Study Part 2 (Part 2a - 0.1% NVC-422, Part 2b - 0.2% NVC-422), once daily for 7 days, held in the bladder for 1 hour
  Other Names: NVC-422

SUMMARY:
The purpose of this clinical trial is to study the effects of NVC-422 instilled into the bladder in reducing bacteria in the urine.

DETAILED DESCRIPTION:
Catheter-associated urinary tract infection (CAUTI) is a major healthcare problem in the U.S., accounting for approximately 40% of all hospital acquired infections. Microorganisms can colonize the catheter extraluminally or intraluminally, and are often protected in a biofilm environment. Nearly all patients catherized for 30 days or longer will develop bacteriuria, or the presence of bacteria in normally sterile urine. Ten to twenty percent of these patients will develop a symptomatic CAUTI. In a further 1-4%, the infection will spread into the kidneys or bloodstream, leading to potentially lethal bacteremia.

Currently, there is no bladder irrigation solution that can reduce or eliminate CAUTI. A bladder instillation solution that can keep the bladder and catheter substantially free of bacteria and biofilm is expected to provide a practical and cost-effective means of minimizing CAUTIs.

NVC-422 is a topical, non-antibiotic, fast acting, broad spectrum anti-microbial, which exhibits potential for the rapid decolonization of a range of urologic pathogens, including Escherichia Coli (E. coli), Enterococcus spp., P. mirabilis and others. In vitro studies with NVC-422 have also shown that it is capable of penetrating a biofilm and effectively killing the contained microbes.

ELIGIBILITY:
Inclusion Criteria:

* Patients or their guardians are willing and able to provide informed consent
* Age > 18 years
* Condition requiring chronic transurethral catheterization for at least 1 month prior to enrollment
* Indwelling transurethral catheter not scheduled for exchange for at least 1 week from first treatment
* Documented asymptomatic bacteriuria as defined in the protocol
* Vital signs within the following limits: blood pressure 90 to 160 mm Hg systolic and 50 to100 mm Hg diastolic, pulse rate 45 to 100 bpm, respiratory rate 8 to 24 respirations per minute, oral body temperature 35.5ºC to 38.0ºC
* Screening must occur within 14 days of enrollment into the study

Exclusion Criteria:

* Unwillingness/inability to fulfill the requirements of the study
* History of hepatitis B or C, HIV, AIDS, or other immunodeficiency disease
* Systemic antibiotics within 7 days of enrollment
* Any condition that, in the opinion of the principal investigator, would make the subject unsuitable for the study or place the subject at additional risk.
* Any investigational drug or investigational device within 30 days of enrollment in the study
* Women who are pregnant or lactating; or of child-bearing potential unless using highly effective birth control method for 1 month prior to and during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-10; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety and antimicrobial effect (and its duration) of NVC-422 in urine following bladder instillation in chronically catheterized subjects with bacteriuria | 7-10 days

SECONDARY OUTCOMES:
Assess urine concentration of NVC-422 and its primary metabolite (2,2-DMT) following bladder instillation | 1-7 days
Assess plasma concentration of NVC-422 and its primary metabolite (2,2-DMT) following bladder instillation | 1-7 days

CONTACTS AND LOCATIONS:
Overall Officials: Rabih O. Darouiche, M.D., Principal Investigator — Baylor College of Medicine
Locations (1):
- Michael E. Debakey V.A. Medical Center, Houston, Texas, United States